CLINICAL TRIAL: NCT01279096
Title: A Phase I Dose Escalation Study of Clofarabine Given in Combination With Multi-agent Therapy for Remission Induction in Pediatric Patients With Acute Lymphoblastic Leukemia in First Relapse or Refractory to First Line Therapy -
Brief Title: Safety of Clofarabine With Multiagent Chemotherapy in Childhood Acute Lymphoblastic Leukemia
Acronym: Vandevol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); Saint-Louis Hospital, Paris, France (Other); Assistance Publique - Hôpitaux de Paris (Other); Hospices Civils de Lyon (Other); University Hospital, Toulouse (Other); Central Hospital, Nancy, France (Other); University Hospital, Marseille (Other); University Hospital, Bordeaux (Other); Nantes University Hospital (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-010826-20; 2008_40/0905 (Other: Sponsor)
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Acute Lymphoid Leukemia Relapse; Acute Lymphoid Leukemia Relapse After Bone Marrow Transplant
Keywords: Acute lymphoblastic leukemia; relapse; childhood; clofarabine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Clofarabine; Etoposide; Asparaginase; Mitoxantrone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Clofarabine — escalating doses of clofarabine starting from 20 mg/m2/day to 40 mg/m2/day from day 1 to day 5 used in association with etoposide, asparaginase, mitoxantrone and dexamethasone
  Other Names: etoposide,; asparaginase,; mitoxantrone; dexamethasone

SUMMARY:
The purpose of this study is to determine Maximum Tolerated Dosage (MTD), Dosage Limited Toxicities (DLT), and the Rate Phase 2 Dosage of clofarabine when used in combination with etoposide, asparaginase, mitoxantrone and dexamethasone and to assess the feasibility and safety of this combination regimen to treat children with high risk relapsed or refractory acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
I.3 Primary Objectives :

To determine the MTD of escalating doses of clofarabine starting from 20 mg/m2/day to 40 mg/m2/day from day 1 to day 5, as a replacement of cytarabine as part of a combination of etoposide, asparaginase, mitoxantrone and dexamethasone (VANDA regimen).

I.4 Secondary Objectives :

1. To determine the safety and tolerability of clofarabine when used in combination with etoposide, asparaginase, mitoxantrone and dexamethasone (VANDA regimen) and determine the duration, seriousness, and relationship of adverse events that occur during the treatment and follow-up periods ; we search DLT
2. To determine the Overall Response rate (OR) (Complete Remission + Complete Remission without platelet's normalization) of clofarabine plus etoposide ,asparaginase, mitoxantrone and dexamethasone (VANDA regimen) in pediatric patients with refractory or relapsed ALL at the established clofarabine RP2D.
3. To document the rate of Partial Response[s] in the study population
4. To document time-to-event parameters, including duration of remission, Event Free Survival (EFS), 4-month EFS, and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* 1 to 21 years old at the date of acute lymphoblastic leukemia initial diagnosis
* Very early medullary first relapse occurring during the first 18th months after complete remission OR patients with second relapse OR a relapse occurring 6 months or more after myeloablative stem cell transplantation will be eligible.
* Have a Karnofsky Performance Status (KPS) of ≥70 for patients >10 years of age or a Lansky Performance Status (LPS) of ≥60 for patients ≤10 years of age.
* No concomitant malignant disease.
* No active uncontrolled infection.
* Have adequate renal and hepatic functions
* absence of concomitant severe cardiovascular disease, i.e. congestive heart failure
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of any investigational agent within 30 days.
* Known hypersensitivity to clofarabine or excipients.
* Known hypersensitivity to mitoxantrone, etoposide or excipients.
* Allergy to both E Coli-Asparaginase and Erwinia Asparaginase
* Prior transplant less than 6 months ago.
* Trisomy 21
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 1 Year to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose of clofarabine in combination with etoposide, asparaginase, mitoxantrone and dexamethasone | within the 40 days after the chemotherapy

SECONDARY OUTCOMES:
efficacy of clofarabine used in combination with etoposide, asparaginase, mitoxantrone and dexamethasone | 40 days after the chemotherapy
  Complete remission rate and minimal residual disease level
Event free survival | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Nelken, MD PhD, Principal Investigator — Lille Unıversity Hospital, Lille, France; Pıerre S Rohrlich, MD, PhD, Study Chair — Besancon University Hospital
Locations (2):
- France (2):
  - Besançon University Hospital, Besançon
  - Lille University Hospital, Lille